CLINICAL TRIAL: NCT07018817
Title: A Trimodal Study on Hypoxia Adaptation: Promotion of Cerebral Functional Connectivity and Decrement of Neuromuscular Efficiency
Brief Title: Hypoxia Adaptation Promotes Cerebral Functional Connectivity With Neuromuscular Efficiency Decrement
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, T.Li, Full professor, Peking Union Medical College
Other Study IDs: Brain Adaptation to Hypoxia
Record Dates: First submitted 2025-04-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-04

CONDITIONS: Hypoxia; Altitude Sickness
Keywords: Brain
MeSH Terms: conditions — Hypoxia; Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: motor execution motor imagery — Participants will perform motor execution tasks and motor imagery tasks following standardized instructions under controlled conditions.

SUMMARY:
The study utilized a trimodal setup comprising EEG, EMG, and fNIRS modules. Participants wore a 64-channel dry EEG cap, while EMG electrodes were placed on the right biceps brachii, the flexor digitorum profundus of the forearm, and the gastrocnemius muscle. fNIRS probes were positioned on the forehead to monitor cerebral hemodynamic responses.

The experimental paradigm included two tasks: motor execution (ME) and motor imagery (MI). During ME, participants performed 15 trials of actual movements. In MI, participants completed 60 trials of imagined movements. Each trial involved a randomly presented stimulus-left-hand clenching, right-hand clenching, or bilateral heel raising-with each movement type occurring an equal number of times across the session.

DETAILED DESCRIPTION:
This study employed a multimodal acquisition system comprising EEG, EMG, and fNIRS modules. Participants were fitted with a 64-channel dry EEG cap for the measurement of cortical electrical activity. Surface EMG electrodes were attached to three muscle groups: the right biceps brachii, the flexor digitorum profundus of the forearm, and the gastrocnemius muscle, to record muscle activation signals. Simultaneously, fNIRS probes were positioned on the participants' foreheads to monitor cerebral hemodynamic responses.

The experimental paradigm was divided into two tasks: motor execution (ME) and motor imagery (MI). During the ME task, participants performed 15 trials of actual movements, whereas the MI task involved 60 trials of imagined movements. Each trial randomly presented one of three stimuli-left-hand clenching, right-hand clenching, or bilateral heel raising-with an equal distribution of the three movement types across the session. The order of stimuli was randomized to prevent prediction bias.

ELIGIBILITY:
Inclusion Criteria:

* People who can withstand altitude sickness

Exclusion Criteria:

* Plateau Native

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Short-term migration from the highlands
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
EEG Power Spectrum in Motor Imagery and Motor Execution Tasks | up to 2 weeks

SECONDARY OUTCOMES:
Surface EMG Amplitude of Upper Limb Muscles during Motor Tasks | up to 2 weeks
Cerebral Oxygenation Measured by Near-Infrared Spectroscopy (NIRS) in Prefrontal Cortex | up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedical engineering，Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.nature.com/articles/s41597-024-03200-8#citeas